CLINICAL TRIAL: NCT04114344
Title: Randomized Clinical Trial to Compare TAPP vs TEP Approach for Women's Inguinal Hernia on an Outpatient Basis
Brief Title: Clinical Trial to Compare TAPP (Transabdominal Preperitoneal) vs TEP (Totally Extraperitoneal) y Approach for Women's Inguinal Hernia on an Outpatient Basis
Acronym: WOLAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, José Tinoco González, Principal Investigator, Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WO_LAP
Record Dates: First submitted 2019-09-12; First posted 2019-10-03 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Inguinal Hernia
Keywords: Woman; Inguinal Hernia; TAPP; TEP; Outpatient Surgery; Ambulatory Surgery
MeSH Terms: conditions — Hernia, Inguinal | interventions — tetra-4-amidinophenoxypropane; tetraethylpyrazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPP (Trans Abdominal PrePeritoneal) (Active Comparator): Trans Abdominal PrePeritoneal approach to inguinal hernia repair
  Interventions: Procedure: TAPP
- TEP (Totally Extra Peritoneal) (Experimental): Totally Extra Peritoneal approach to inguinal hernia repair
  Interventions: Procedure: TEP

INTERVENTIONS:
Procedure: TAPP — Trans Abdominal Pre Peritoneal approach
  Arms: TAPP (Trans Abdominal PrePeritoneal)
Procedure: TEP — Total Extra Peritoneal approach
  Arms: TEP (Totally Extra Peritoneal)

SUMMARY:
Open prospective randomised clinical trial enrolling women who suffer from inguinal or femoral hernia, to evaluate if TEP approach is superior to TAPP concerning postoperative development, principally postoperative pain, with no increase of recurrent hernia at the one-year follow-up visit.

DETAILED DESCRIPTION:
Randomised phase IV clinical trial enrolling women suffering from inguinal hernia in Virgen del Rocío University Hospital influence area, from March 2019 to March 2021.

The aim of the study is to conclusively stablish whether there is real and significant benefit in using TEP approach over TAPP, in an outpatient basis, concerning postoperative evolution. Secondary objectives are the assessment of postoperative pain, using VAS (visual analogic scale), of both techniques, and evaluation of hernia recurrence during the first postoperative year The individuals will be assigned to each group according to simple random sampling.

ELIGIBILITY:
Inclusion Criteria:

* Inguinofemoral hernia, EHS (European Hernia Society) classification.
* Patient over 18 years old.
* Signed informed consent form.
* Female
* Meeting of outpatient discharge criteria, determined by Aldrete´s test

Exclusion Criteria:

* Loss of domain.
* Abdominal skin grafts.
* Previous preperitoneal (open or laparoscopic) prosthetic mesh.
* Incarcerated hernia.
* Previous complications such as infection, fistulae…
* Not candidate for ambulatory surgery
* Pregnancy or desire for pregnancy in the first postoperative year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 24 hours
  Post operative pain, measured with Visual Analogue Scale (VAS) (from 0 to 10 points) World Health Organization (WHO)
Recurrence | One year
  Recurrence of inguinal hernia in the one-year follow-up
Complications | One year
  Postoperative complications including wound complications (seroma, haematoma, infection), gastrointestinal complications (ileus, fistula), urological complications (acute retention, haematuria) and hernia complications (recurrence, chronic groin pain) will be reported. Occurrence of major complications will be registered, including intestinal injury, major vascular lesion, bleeding over 500cc and peritonitis.

SECONDARY OUTCOMES:
Operating time | 180 minutes
  Operating time from first incision to closure
Hospital stay | 24 hours
  length of hospital stay will be measured in hours between the end of the surgery and the time of discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Virgen del Rocío University Hospital, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT04114344/ICF_000.pdf